CLINICAL TRIAL: NCT04382638
Title: Effectiveness of Three Dimensional Correction During in Bracing in Adolescent Idiopathic Scoliosis: a Prospective Randomised Clinical Trial of Rigo Chêneau Versus Boston-style Orthoses
Brief Title: Effectiveness of Three Dimensional Correction During in Bracing in Adolescent Idiopathic Scoliosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The University of Hong Kong (Other)
Collaborators: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Kenny Kwan, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UW 20-243
Record Dates: First submitted 2020-05-05; First posted 2020-05-11 (Actual); Last update posted 2023-02-06 (Actual); Status verified 2023-02

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: AIS

STUDY DESIGN:
Intervention Model Description: Patients diagnosed with AIS referred for bracing through the hospital's specialist outpatient clinic are eligible to enrol the study. The Investigator will document whether each patient meets the selection criteria before enrolment into the study. The Investigator or designee will also obtain an IRB/EC approved Informed consent from each patient and/or guardian.
  Eligible patients will be randomly assigned to either RCO group (experimental) or TLSO group (control) in a ratio of 1:1. The radiographic evaluation, physical examination and PROM questionnaires will be assessed at baseline, 3 months, 6 months, 12 months and every year until patients reach skeletal maturity or if surgical intervention is required.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Assessor, statistician and investigator blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RCO group (Experimental): Patients in the experimental group will receive RCO fabrication with standard level of care for bracing, which consists of education on general exercises for spinal movement, strengthening, and balancing. These patients will attend study assessments at baseline, 3 months, 6 months, 12 months and every year until they reach skeletal maturity or if surgical intervention is required.
  Interventions: Combination Product: RCO group
- TLSO group (Active Comparator): Patients in the experimental group will receive TLSO fabrication with standard level of care for bracing, which consists of education on general exercises for spinal movement, strengthening, and balancing. These patients will attend study assessments at baseline, 3 months, 6 months, 12 months and every year until they reach skeletal maturity or if surgical intervention is required.
  Interventions: Device: TLSO group

INTERVENTIONS:
Combination Product: RCO group — Patients in the experimental group will receive RCO fabrication with standard level of care for bracing, which consists of education on general exercises for spinal movement, strengthening, and balancing. These patients will attend study assessments at baseline, 3 months, 6 months, 12 months and every year until they reach skeletal maturity or if surgical intervention is required.
  Arms: RCO group
Device: TLSO group — Patients in the experimental group will receive TLSO fabrication with standard level of care for bracing, which consists of education on general exercises for spinal movement, strengthening, and balancing. These patients will attend study assessments at baseline, 3 months, 6 months, 12 months and every year until they reach skeletal maturity or if surgical intervention is required.
  Arms: TLSO group

SUMMARY:
The purpose of this study is to study the effectiveness of in-brace 3D scoliosis correction by comparing Rigo Chêneau orthoses (RCO) with conventional Traditional Boston-style thoracolumbosacral orthoses (TLSO) in Adolescent Idiopathic Scoliosis (AIS) patients, following Scoliosis Research Society (SRS) and The International Scientific Society on Scoliosis Orthopaedic and Rehabilitation Treatment (SOSORT) recommendations for non-operative AIS management and research studies. This group of patients that reach the threshold for bracing have an intrinsic higher risk for curve progression. Hence, the proposed study will provide novel and high quality evidence to improve the efficacy of bracing in the non-operative treatment of AIS. This will contribute significantly to the betterment of public health by reducing the number of patients requiring surgical intervention. Ultimately, new evidence-based clinical practice guidelines on the most effective type of scoliosis braces will benefit children diagnosed with AIS worldwide.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS), a three-dimensional (3D) deformity of the spinal column characterized by lateral deviation and vertebral rotation, affects 3.5% of children during puberty in Hong Kong. Untreated scoliosis continues to deteriorate beyond adolescence, and curves that progress beyond 50 degrees can lead to chronic back pain, cardiopulmonary compromise, poor cosmesis and negative psychological impact. Hence, surgical correction of the deformity by instrumented spinal fusion is recommended when curves reach 50 degrees. Although surgical risks have decreased with improved techniques, surgeries for scoliosis correction still carry significant medical co-morbidities, psychological stress to the children and their families, and substantial financial burden on healthcare. Effective non-operative strategies to prevent curve progression during adolescence are needed. Currently, the most effective non-operative treatment supported by high quality randomised controlled trial to prevent curve progression is by spinal bracing. In the Bracing in Adolescent Idiopathic Scoliosis Trial (BrAIST) study, bracing was effective in preventing curve progression to threshold for surgery in 72% of cases. The failure rate, therefore, remains substantially high despite the best available non-operative treatment. Previous studies have identified factors affecting brace success, including skeletal age, curve type, curve magnitude, and flexibility, but none of these is modifiable. Brace treatment requires a wholistic approach, and brace design and fabrication are important determinants of brace effectiveness. Traditional Boston-style thoracolumbosacral orthoses (TLSO), such as those used in the BrAIST study, can achieve in-brace coronal curve correction reliably but their effects on the 3D curve correction are highly variable. Since AIS is a 3D deformity, it is reasonable to postulate that braces which can achieve correction in all three planes have a higher chance of success.

Rigo Chêneau orthoses (RCO) were developed approximately two decades ago by Dr. Manuel Rigo of Barcelona who made improvements to the Chêneau brace that French doctor Jacques Chêneau invented in 1978. RCO was designed with the intent to combine biomechanical forces in three dimensions, including curve derotation. They use an open pelvis design with anterior opening. Instead of focusing on one-dimensional correction, RCO treats scoliosis in all three dimensions and follows a unique curve Rigo classification protocol to guide brace design. RCO not only keeps the curves from getting worse as seen on an X-ray, but also corrects as much as possible the way the body looks. Every attempt is made to decrease the noticeable effects of scoliosis such as rib humps, uneven shoulders, hips which are translated or rotated, and centering the head over the pelvis. To achieve successful 3D scoliosis correction, in-brace Cobb angle correction must be 50% to be considered acceptable. This is often true and it is also true that the Cobb angle, which is easily assessed, has been the gold standard of measurement for brace quality. However, not all patients can and/or should be corrected to 50% in-brace correction. In some cases, a 25% in-brace correction coupled with good 3D correction is acceptable and sufficient to prevent scoliosis progression, when greater Cobb angle correction would cause negative compensations. Overall, some patients are best served by targeting a low in-brace correction, whereas for others an 80% in-brace correction is both achievable and desirable.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of AIS
* Male or female from 10 to 15 year-old, inclusive, at the time of consent provided
* Skeletal immaturity, defined as a Risser grade (amount of ossification and eventual fusion of the iliac apophysis) of 0, 1, or 2
* Cobb angle of 25-40
* No prior conservative or surgical treatment for AIS

Exclusion Criteria:

* An underlying cause or association that may cause scoliosis
* Leg length discrepancies or lower limb deformities that may interfere with spinal posture
* Previous spinal surgery
* Cognitive impairment
* Those receiving any other forms of treatment including alternative medicine for the treatment of their scoliosis
* Those who are unable to return for follow-up to complete the trial

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 134 (Estimated)
Dates: Start 2022-07-02 (Actual); Primary Completion 2025-07-03 (Estimated); Study Completion 2025-12-03 (Estimated)

PRIMARY OUTCOMES:
Effect of in-brace 3D scoliosis correction between RCO versus TLSO as determined by the difference in coronal Cobb angle pre- and one year post-treatment | baseline, 3 months, 6 months, 12 months up to 5 years
  To evaluate the effect of in-brace 3D scoliosis correction between RCO versus TLSO as determined by the difference in coronal Cobb angle pre- and one year post-treatment

SECONDARY OUTCOMES:
Compare changes in sagittal plane radiological parameter between RCO versus TLSO by EOS Imaging System | baseline, 3 months, 6 months, 12 months up to 5 years
  To evaluate the effect of in-brace 3D scoliosis correction between RCO versus TLSO on sagittal plane radiological parameter using EOS Imaging System
Compare changes in transverse plane radiological parameter between RCO versus TLSO by EOS Imaging System | baseline, 3 months, 6 months, 12 months up to 5 years
  To evaluate the effect of in-brace 3D scoliosis correction between RCO versus TLSO on transverse plane radiological parameter using EOS Imaging System
Compare changes in surface topography between RCO versus TLSO using Bunnell's scoliometer | baseline, 3 months, 6 months, 12 months up to 5 years
  To evaluate the effect of RCO during in-bracing on surface topography using Bunnell's scoliometer with a range from 0 degree to 30 degree (left/right). Reading closer to 0 degree indicates better surface topography
Compare changes in surface topography between RCO versus TLSO using clinical photography | baseline, 6 months, 12 months up to 5 years
  To evaluate the effect of RCO during in-bracing on surface topography using clinical photography
Compare changes in surface topography between RCO versus TLSO using VITUS Smart XXL 3D body scanner system | baseline, 6 months, 12 months up to 5 years
  To evaluate the effect of RCO during in-bracing on surface topography using VITUS Smart XXL 3D body scanner system
Measure changes in quality of life between RCO versus TLSO by Scoliosis Research Society-7 questionnaire | baseline, 6 months, 12 months up to 5 years
  To measure changes in quality of life between RCO versus TLSO by Scoliosis Research Society-7 questionnaire, with the minimum score of 22 to the maximum score of 110. Higher score indicates better health outcome
Measure changes in health outcome between RCO versus TLSO by EQ-5D-5L | baseline, 6 months, 12 months up to 5 years
  To measure changes in health outcome between RCO versus TLSO by EQ-5D-5L, with the part of EQ-VAS score ranging from the minimum of 0 to the maximum of 100. Higher score indicates better health outcome
Measure changes in patients' perception of their appearance between RCO versus TLSO by Trunk Appearance Perception Scale | baseline, 6 months, 12 months up to 5 years
  To measure changes in patients' perception of their appearance between RCO versus TLSO by Trunk Appearance Perception Scale with 5 graphical illustrations. Graph 1 represents the patient's best self-perception of his or her appearance while graph 5 represents the patient's worst self-perception of his or her appearance
Measure changes in levels of pain between RCO versus TLSO by Numeric Pain Ratings | baseline, 6 months, 12 months up to 5 years
  To measure changes in levels of pain between RCO versus TLSO by Numeric Pain Ratings with a range from the minimum of 0 to the maximum of 10. Lower score indicates less pain.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kenny Kwan, BMBCh (Oxon), Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No